CLINICAL TRIAL: NCT05218811
Title: Cryotherapy and Robotic Assisted Non Ischemic Nephron Sparring Surgery
Brief Title: Cryaoablation Assisted Partial Nephrectomy a Non Ischemic Approach
Acronym: RCAPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urological Research Network, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URN-202000244
Record Dates: First submitted 2021-09-26; First posted 2022-02-01 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are scheduled for a surgical procedure: robotic partial nephrectomy, and the investigators will use a cryoablation probe(s) for selective ischemia rather than full blood flow interruption with a vascular clamp
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental): Patients underwent Cryotheapy assisted partial nephrectomy
  Interventions: Device: Cryoablation Assisted Partial Nephrectomy

INTERVENTIONS:
Device: Cryoablation Assisted Partial Nephrectomy — Cryoablation Assisted Partial Nephrectomy is monitored under Ultrasound guidance, A Cryoablation machine (FDA Approved Device) along with its Cryoprobes are used in the study The Cryoprobes are placed in close to the endophytic tumor margins. The tumor boundary area will undergo one freezing cycles. Tumor is excised after 5 minutes of freezing cycle. Thawing process is passive, renal defect repair is conducted during thawing process.

SUMMARY:
Patients with renal masses eligible to partial nephrectomy often require arterial ischemia to control or prevent blood loss during this surgical procedure. This study aims to determine the safety and efficacy of renal cryoablation at the tumor bed, as a substitute measure or technique vs total or selective arterial renal ischemia.

DETAILED DESCRIPTION:
Nephron sparring surgery has emerged as the procedure of choice for most patients with renal tumors that are >2 cm and harbor a greater than 50% exophitic component. In order to decrease blood loss surgeons may: 1- interrupt blood flow to the kidney, completely or selectively; 2-Use diuretics such as mannitol to dehydrate the kidney; 3-Ice externally the kidney - in open procedures - to decrease metabolism during ischemia.

The emergence of robotic surgery triggered a shift in the the surgical approach to partial nephrectomy and is commonly employed. A fundamental drawback of this technique is represented on the lack of cold ischemia. However, warm ischemia is commonly employed and requires dissection of the renal pedicle, which by itself puts the kidney at risk of loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ages between 45-90-year-old.
* Renal tumor ≤ 7 cm in the greatest extension, >50% exophitic.

Exclusion Criteria:

* Prior renal surgery
* M1 Disease

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2041-05-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence - Oncological Control | 10 Years
  Recurrence at Site of Excision or within 1 cm of margin or Development of Metastasis

SECONDARY OUTCOMES:
Local Re-Intervention | 10 Years
  Either subsequent ablation or surgical exploration or surgical kidney removal
Development or Progression of Chronic Kidney Disease (CKD) | 10 Years
  De-Novo emergence of CDK or changes in CKD overtime based on variation from baseline. The international classification for CKD defined by serum estimated Glomerular Filtration Rates (GFR) will be used as measurement instrument using the following definitions:
  GFR categories in CKD G1 ≥90 Normal or high G2 60-89 Mildly decreased* G3a 45-59 Mildly to moderately decreased G3b 30-44 Moderately to severely decreased
Incidence of Metastatic disease | 10 Years
  patients will be evaluated using imaging studies at fixed intervals as follows: at 6 months Renal Ultrasound at 1 year CT Urogram at 18 Months, 24 months and yearly thereafter with Renal Ultrasound CT Urograms will be performed as needed for cause
Survival | 10 years
  If a patient expiries during the study interval we would procure the death certificate and do our best to determine cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Bianco, MD, Principal Investigator — Urological research Network
Locations (1):
- Urological Research Network, Miami Lakes, Florida, United States

REFERENCES:
- [Background] Ismail M, Nielsen TK, Lagerveld B, Garnon J, Breen D, King A, van Strijen M, Keeley FX Jr. Renal cryoablation: Multidisciplinary, collaborative and perspective approach. Cryobiology. 2018 Aug;83:90-94. doi: 10.1016/j.cryobiol.2018.06.002. Epub 2018 Jun 8. PMID 29890126
- [Background] Makki A, Aastrup MB, Vinter H, Ginnerup B, Graumann O, Borre M, Nielsen TK. Renal cryoablation - does deep endophytic ablation affect the renal collecting system? Scand J Urol. 2020 Feb;54(1):33-39. doi: 10.1080/21681805.2019.1702094. Epub 2019 Dec 16. PMID 31842655
- [Background] Berger A, Kamoi K, Gill IS, Aron M. Cryoablation for renal tumors: current status. Curr Opin Urol. 2009 Mar;19(2):138-42. doi: 10.1097/MOU.0b013e328323f618. PMID 19188767
- [Background] Ushijima Y, Asayama Y, Nishie A, Takayama Y, Kubo Y, Ishimatsu K, Ishigami K. Cryoablation for Secondary Renal Cell Carcinoma After Surgical Nephrectomy. Cardiovasc Intervent Radiol. 2021 Mar;44(3):414-420. doi: 10.1007/s00270-020-02709-w. Epub 2020 Nov 17. PMID 33205290
- [Background] Zargar H, Atwell TD, Cadeddu JA, de la Rosette JJ, Janetschek G, Kaouk JH, Matin SF, Polascik TJ, Zargar-Shoshtari K, Thompson RH. Cryoablation for Small Renal Masses: Selection Criteria, Complications, and Functional and Oncologic Results. Eur Urol. 2016 Jan;69(1):116-28. doi: 10.1016/j.eururo.2015.03.027. Epub 2015 Mar 26. PMID 25819723